CLINICAL TRIAL: NCT05714020
Title: Effects of High-frequency RTMS on Brain Connectivity
Brief Title: TMS-evoked Potentials During Repetitive Transcranial Magnetic Stimulation on the Primary Motor Cortex
Acronym: rTMS-TMS-EEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Enrico De Martino, Principal Investigator, Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20220018-1
Record Dates: First submitted 2023-01-25; First posted 2023-02-06 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Repetitive Transcranial Magnetic Stimulation; Motor Cortex; Transcranial Magnetic Stimulation; Pain Thresholds; Electroencephalography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Real rTMS (Active Comparator): The active rTMS protocol is a 15-minute 10Hz stimulation, 10 seconds on, 20 seconds off, at 90% RMT, for a total of 3000 pulses using a real TMS coil. The target is the primary motor cortex.
  Interventions: Other: Real rTMS
- Sham rTMS (Sham Comparator): The sham rTMS protocol is performed by a sham coil. The sham rTMS protocol is a 15-minute 10Hz stimulation, 10 seconds on, 20 seconds off, at 90% RMT, for a total of 3000 pulses. The target is the primary motor cortex.
  Interventions: Other: Sham rTMS

INTERVENTIONS:
Other: Real rTMS — Repetitive transcranial magnetic stimulation (rTMS) is applied to the primary motor cortex. The protocol consists of 15 minutes of 10Hz stimulation, 10 seconds on, 20 seconds off, at 90% RMT, for a total of 3000 pulses.
  Arms: Real rTMS
Other: Sham rTMS — A sham coil is also used to mimic the clicking sound of the transcranial magnetic coil and skin stimulation.
  Arms: Sham rTMS

SUMMARY:
This study investigates the modification of the local-to-global connectivity pattern in response to a session of repetitive transcranial magnetic stimulation (rTMS) applied to the primary motor cortex. Transcranial magnetic stimulation (TMS) will be applied to elicit electroencephalography (EEG) responses in healthy volunteers. The TMS-evoked potentials (TEPs) will be recorded and serve as a reflection of cortical reactivity to TMS.

DETAILED DESCRIPTION:
Abnormal connectivity patterns interfere with the normal function of a given neuronal network, thus leading to circuit dysfunction and, subsequently, chronic pain. In the last few years, neuroscience has been heavily influenced by network science. This synergistic association provided a new framework for understanding brain function in health and how dysfunction in specific neuronal brain circuits can lead to symptoms. A network comprises nodes (e.g., areas of the brain) and edges (functional connections between nodes). An effective network can process and share large amounts of information while maintaining specificity and not allowing noise to contaminate the flow of information across the circuits. The network approach to brain functioning has been able to integrate what has been known for several decades as spatial structural anatomy with the time-varying streaming of information (connectivity) in a dynamic perspective. In this context, symptoms of diseases are seen as being correlated with specific network abnormalities, and therapeutic interventions as being associated with the normalisation of these abnormal patterns of connection. Non-invasive neuromodulatory approaches, such as repetitive transcranial magnetic stimulation (rTMS), have entered the guidelines for the management of major depression refractory to pharmacological treatment (FDA clearance in 2008 - K061053) and several chronic pain conditions, providing low-adverse event, rapid-to-perform and safe non-pharmacological treatment possibilities for neuropsychiatric disorders. rTMS is based on the induction of a high-intensity magnetic field on the scalp and on the subsequent creation of an induced electric current that penetrates the skull and influences neuronal firing over a very restricted volume of the brain. Depending on stimulation parameters, rTMS also acts by facilitating or depressing the activity of specific brain networks non-invasively. Despite important advances in the use of rTMS, and similar to what is also obtained from pharmacological treatments, up to 40% of patients remain symptomatic after treatment. This study aims to investigate the responses of specific neuronal brain circuits to repetitive transcranial magnetic stimulation (rTMS) applied to the primary motor cortex in healthy volunteers. It has been hypothesised that the local-to-global connectivity pattern obtained by the stimulation of different cortical hubs (primary motor cortex, dorsolateral prefrontal cortex, anterior cingulate cortex and posterior insula) will be described by TMS-EEG responses in healthy individuals. The modification in cortical connectivity in response to a repetitive transcranial magnetic stimulation (rTMS) applied to the primary motor cortex will be described and compared with a sham rTMS stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Speak and understand English

Exclusion Criteria:

* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous neurologic, musculoskeletal or mental illnesses
* Lack of ability to cooperate
* History of chronic pain or current acute pain
* Contraindications to rTMS application (history of epilepsy, metal in the head or jaw etc.).
* Failure to pass the "TASS questionnaire" (TASS = Transcranial Magnetic Stimulation Adult Safety Screen)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Cortical connectivity | Cortical connectivity changes will be investigated before and after rTMS (1 hour)
  Global and local mean field amplitude

SECONDARY OUTCOMES:
Cortical excitability | Cortical excitability changes will be investigated before and after rTMS (1 hour)
  TMS-evoked potentials

CONTACTS AND LOCATIONS:
Overall Officials: Enrico De Martino, MD, PhD, Principal Investigator — Aalborg University
Locations (1):
- Aalborg University, Gistrup, North Denmark, Denmark